CLINICAL TRIAL: NCT01201993
Title: Observational Study Following After Patients Admitted With Syncope
Brief Title: Clinical and Laboratory Characteristics of Patients Admitted With Syncope; Diagnosis and Follow up After These Patients
Status: Suspended | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: George S. Habib, Dept of Medicine, Carmel Medical Center
Other Study IDs: SYN2010
Record Dates: First submitted 2010-08-17; First posted 2010-09-15 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2010-09

CONDITIONS: Diagnosis; Recurrence
Keywords: syncope; evaluation; recurrence; morbidity
MeSH Terms: conditions — Disease; Recurrence; Syncope

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators hypothesis is that a significant number of patients may remain without specific cause and have recurrent syncope with its associated physical and mental morbidity.

DETAILED DESCRIPTION:
1. Patients with diagnosis of syncope who were admitted to the medical ward will be interviewed and their charts reviewed to rule in or out the diagnosis of syncope.
2. Assess physical and mental injury as a result of syncope.
3. The lab workup will be documented including;

   1. - Routine blood tests.

      * troponin level.
   2. - ECG.

      * Echocardiogram
      * Brain CT.
      * EEG.
      * U/S doppler of carotids.
      * Tilt tests.
4. At the time of diagnosis the final diagnosis will be documented including recommendations for patients to prevent syncope after discharge.
5. Follow up after patients by phone verifying recurrence of syncope and resulting physical and or mental injury if any.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosis of syncope on admission to the medical ward.

Exclusion Criteria:

* patients with loss of consciousness due to other than low perfusion of the brain
* patients that can't sign a consent form
* patients that we can't get details about the episode of the syncope

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted patients the medical ward
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-08; Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
diagnosis | 1 year
  Final diagnosis as a cause of syncope

SECONDARY OUTCOMES:
recurrence | 6 months
  how many patients had recurrence of syncope and average number of syncope in these patients during the period of follow up of each patient.
physical injury | 6 months
  During this period of follow up of each patient, was there a physical injury, graded either none, mild, moderate or severe (bedridden)
Mental effect | 6 months
  fear of recurrent syncope affecting his mobility and graded from mild to severe where severe indicates fear of moving even one step without support.

CONTACTS AND LOCATIONS:
Overall Officials: George S Habib, M.D., Principal Investigator — Carmel Medical Center
Locations (1):
- Department of Medicine, Carmel Medical Center, Haifa, Israel